CLINICAL TRIAL: NCT06071065
Title: Impact of Clinical Pharmacist Intervention on Medication Adherence and Its Association with Clinical Outcomes in Chronic Kidney Disease in Islamabad
Brief Title: Clinical Pharmacist Intervention on Medication Adherence and Clinical Outcomes in Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Matti Ullah, Assistant Professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU0823-IS
Record Dates: First submitted 2023-09-20; First posted 2023-10-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease
Keywords: Clinical Pharmacist Intervention; Medication Adherence; Clinical outcomes; Health related Quality of life
MeSH Terms: conditions — Renal Insufficiency, Chronic; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were not informed of which groups they belonged to and what type of intervention is provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic (Active Comparator): Basic intervention included the usual counselling by a clinical pharmacist e.g.
  1. Patients Education
     * Pharmacist counseling regarding their disease type and severity
     * Pharmacist counseling (15- to 20-minute sessions) on the proper use of medication
     * Pharmacist counseling regarding the importance of their therapy (treatment)
     * Labeling of medication packs to assist pill sorting. Labels included instructions on dose and frequency/ timing of medication doses
  2. Optimizing therapy monitoring
     * Prescription information quality (incomplete prescription)
     * wrong dose
     * wrong frequency etc.
  Interventions: Behavioral: Pharmacist counselling
- Advanced (Experimental): In addition to Basic Intervention:
  1. Preventing drug interactions :
     • Detection or assessment of potential DDIs by a pharmacist prior to the start of treatment and recommendations for their management.
  2. Patient Education regarding Medications :
     * Pharmacist counseling (15- to 20-minute sessions) on the proper use of medication.
     * Pharmacist counseling on the safe use of medication (self-medication or over-the-counter [OTC] medicines)
  3. Preventing an adverse drug event
     • Monitoring, and prompt detection of adverse drug events (ADEs)
  4. Education on lifestyle modifications
     * Education on lifestyle e.g. regarding exercise
     * Renal diet plan will be given to patients
  5. Renal Dose Adjustments :
     * Detection or assessment of potential nephrotoxic drugs by a pharmacist prior to start of treatment and recommendations for their renal dose adjustment.
  Interventions: Behavioral: Pharmacist counselling

INTERVENTIONS:
Behavioral: Pharmacist counselling — Counselling session with Pharmacist about disease and medication therapy.

SUMMARY:
The purpose of this research study is to evaluate the impact of clinical pharmacist interventions on treatment outcomes, health-related quality of life (HRQoL),and medication adherence among chronic kidney disease patients.

Pharmacist's intervention aim to answer:

1. How a clinical pharmacist intervention program impact medication adherence in chronic kidney disease?
2. To assess how patients' counseling and medication adherence impact patient health-related quality of life?
3. How a clinical pharmacist intervention program improves clinical outcomes of chronic kidney disease patients?

DETAILED DESCRIPTION:
This is a randomized, pharmacist-led, two-group, longitudinal descriptive intervention study performed at a private hospital nephrology department. The study included the introduction of clinical pharmacist interventions to improve adherence to prescribed medications, health-related quality of life, and clinical outcomes in patients with Chronic Kidney Disease(CKD).

Recruited patients were randomly divided into two groups; the basic intervention group and the advanced intervention group.

The basic intervention group received routine counseling. An advance intervention group was provided in addition to the usual counseling, education about Chronic Kidney Disease, hypertension or other comorbidity and management, as well as medication adherence, and renal diet (educational infographic for Chronic Kidney Disease patients) at three follow-up intervals after every 2 months. Both groups were followed up for a period of 6 months.

Pre-validated questionnaires will be used for the assessment

1. Medication Adherence Rating Scale (MARS): to evaluate medication adherence
2. MOS 36-Item Short Form Survey Instrument (SF-36): For evaluation of health related quality of life.

For evaluation of clinical outcome Blood pressure, serum creatinine, and hemoglobin will be obtained from medical records (from hospital software or from patient who had done their labs from out sources)during the baseline visit. The same laboratory tests will also be assessed at patients three-time intervals at admission or first visit at the start of treatment, week 8, and week 16.

ELIGIBILITY:
Inclusion Criteria:

* All male and female inpatients and outpatients with chronic kidney disease defined as a creatinine clearance (CrCl) less than 60 ml/min/l, 73 m2
* over the age of 18 years , will be included in study.
* Patient who are on maintenance hemodialysis also included.

Exclusion Criteria:

* Patients with acute renal failure
* Patients who are receiving renal transplants will not be included.
* Patients who will refuse to participate in study will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Health related Quality of Life | 6 months
  Patients health related quality of life will be assessed using pre-validated tool RAND-36
Patients Medication Adherence. | 6 months
  The primary aim of this study will be to evaluate the effectiveness/impact of a clinical pharmacist intervention program on medication adherence in chronic kidney disease.
  Adherence will be measured using Medication Adherence Repoting Scale (MARS-10). This scale describes three-dimension ,medication adherence behaviour (1-4),attitude towards taking medication (5-8),negative side effects and attitudes to psychotropic medication (9-10).
  Each question has Yes and No response, a response with medication adherence coded as 1 and with non-adherence coded as 0. higher the score higher will be adherence and vice versa.score <6 showes poor adherence and > 8 showes good adherehnce.

SECONDARY OUTCOMES:
Serum Creatinine | 6 months
  Change in serum creatinine levels after intervention
Blood Pressure | 6 months
  Change in Mean arterial Blood pressure
Haemoglobin | 6 months
  Change in blood haemoglobin levels following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Matti Ullah, PhD, Study Director — Hamdard University Islamabad Campus; Iqra Sagheer, Principal Investigator — Akbar Niazi Teaching Hospital; Muhammad Masoom Akhter, PhD, Study Chair — Hamdard University Islamabad Campus
Locations (1):
- Akbar Niazi Teaching Hospital, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Depends on the patient Consent